CLINICAL TRIAL: NCT04104646
Title: A Phase II, Multicenter, Double Blind, Double Dummy, Randomized, 2 Arms Parallel Study to Evaluate the Efficacy, Safety and Pharmacokinetics of CHF6563 in Babies With Neonatal Opioid Withdrawal Syndrome
Brief Title: CHF6563 in Babies With Neonatal Opioid Withdrawal Syndrome
Acronym: NOWSHINE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLI-06563AA1-02
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Opioid Withdrawal Syndrome
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind, double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CHF6563 (Experimental): Sublingual dose of CHF6563 and the corresponding oral dose of morphine matched placebo
  Interventions: Drug: CHF6563; Drug: Morphine matched placebo
- Morphine (Active Comparator): Oral dose of morphine and the corresponding sublingual dose of CHF6563 matched placebo.
  Interventions: Drug: Morphine; Drug: CHF6563 matched placebo

INTERVENTIONS:
Drug: CHF6563 — Sublingual CHF6563 administration at starting dose of 10 µg/kg q8
  Arms: CHF6563
Drug: Morphine — Oral morphine administration at starting dose of 0.07 mg/kg q4
  Arms: Morphine
Drug: CHF6563 matched placebo — Sublingual CHF6563 matched placebo administration
  Arms: Morphine
Drug: Morphine matched placebo — Oral morphine matched placebo administration
  Arms: CHF6563

SUMMARY:
A Phase II, multicenter, double blind, double dummy, randomized, 2 arms parallel study to evaluate the efficacy, safety and pharmacokinetics of CHF6563 in babies with Neonatal Opioid Withdrawal Syndrome

DETAILED DESCRIPTION:
This was a randomised, multicentre, double-blind, double-dummy, parallel-group, controlled study of CHF6563 (non-ethanolic buprenorphine) sublingual solution.

For the enrolled subjects, withdrawal signs were assessed using a pre-defined Finnegan Neonatal Abstinence Scoring Tool (FNAST). FNAST assessments were made in neonates who showed signs of withdrawal despite appropriate non-pharmacological care and were recorded every 4 hours (±1 hour). Pharmacological treatment was to be started up to 7 days after birth in neonates who showed signs of neonatal opioid withdrawal syndrome (NOWS), defined as the sum of three consecutive FNAST scores ≥24 or a single score ≥12, and had failed to respond to non-pharmacological care. After FNAST assessment had started, it was continued for at least 24 hours, even if the baby was not randomised.

Sublingual administration of CHF6563 (non-ethanolic buprenorphine) solution (0.075 mg/mL) at a starting dose of 10 μg/kg every 8 hours (q8), using birth weight and oral administration of morphine-matched placebo (sterile water for injection USP), every 4 hours (q4). Thereafter, up-titrations of CHF6563 were possible to a maximum scheduled dose of 90 μg/kg/day. At the discretion of the physician, rescue doses of CHF6563 or morphine could have been given during the treatment to a neonate who had a single score of ≥12. Duration of treatment could last a maximum of 10 weeks. Adverse events (AEs) and serious adverse events (SAEs) were collected starting from the time of informed consent signature or from the neonate's birth (if the informed consent was signed before birth) through treatment and the follow-up period.

The study was terminated for non-safety reasons on 04 February 2022, due to low recruitment rate, after only 7 subjects out of a planned 57 subjects had been randomised. An Independent Safety Monitoring Board (ISMB) was in-place to review the safety profile of CHF6563/morphine treatment; the study was terminated before the ISMB reviewed any data.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained by parents/legal representative(according to local regulation) prior to or after birth.
2. Birth weight ≥ 3rd centile for gestational age (GA), according to the Centers for Disease Control and Prevention (CDC) growth chart
3. Gestational age ≥ 36 weeks
4. Exposure to opioids during the last month of fetal life
5. Signs of neonatal opioid withdrawal syndrome requiring treatment, and the sum of 3 consecutive FNAST scores is ≥ 24 or a single score ≥ 12

Exclusion Criteria:

1. Familial history of prolonged QTc syndrome
2. Major congenital malformations or evidence of congenital infection
3. Signs of fetal alcohol spectrum disorders
4. Maternal alcohol abuse, defined as average of 3 or more drinks per week in the last 30 days
5. Medical illness at the time of randomization, including but not exclusively:

   1. Neonatal hypoglycemia requiring intravenous glucose therapy
   2. Neonatal respiratory illness requiring non-invasive or invasive respiratory support
   3. Neonatal encephalopathy (including hypoxic ischemic encephalopathy or seizures
   4. Severe hyperbilirubinemia-bilirubin at or above the exchange transfusion threshold as defined by the American Academy of Pediatrics (AAP)
   5. Severe elevation of serum aminotransferases (more than twice the upper limit of the age appropriate aminotransferases reference range of the investigational site).
   6. Proven or suspected early onset neonatal infection which will require more than 48 hours treatment with antibiotics
6. Unable to tolerate an oral or sublingual medication
7. Need for medications forbidden in this study protocol
8. Any condition that, in the opinion of the Investigator, would place the neonate at undue risk
9. Participation in another clinical trial of any medicinal product, placebo, experimental medical device or biological substance conducted under the provisions of a protocol on the same therapeutic target. The participation in studies involving diagnostic devices or treatments for conditions other than NOWS and Neonatal abstinence syndrome (NAS) may be permitted following an agreement with the Sponsor. Non-interventional observational studies are allowed

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kraft, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Clinical site 015, Las Vegas, Nevada
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHF6563 | Morphine
Started | 5 | 2
Completed | 1 | 1
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHF6563 | Morphine | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: days] | 1.0 (0.7) | 0.5 (0.7) | 0.9 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 2 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7
Gestational age [Mean (Standard Deviation); unit: weeks] | 38.37 (1.17) | 39.14 (1.62) | 38.59 (1.22)
Body length [Mean (Standard Deviation); unit: cm] | 49.16 (2.37) | 50.90 (0.14) | 49.66 (2.12)
Weight [Mean (Standard Deviation); unit: kg] | 3.1718 (0.5319) | 3.7980 (0.8669) | 3.3507 (0.6382)
Head circumference [Mean (Standard Deviation); unit: cm] | 33.50 (1.12) | 35.50 (2.12) | 34.07 (1.59)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Treatment
Description: Duration of treatment defined as the number of hours from first dose of study drug administration until the last dose of study drug.
  Shown are results for the duration of treatment in all treated patients, regardless of discontinuation status, as well as those patients who completed the study (with non missing data).
  The number of subjects randomised in the study was much lower than planned. Although data from 5 subjects were used in the CHF6563 treatment group, only 2 subjects completed the study as planned i.e. 1 subject in each study arm; no imputation of missing or incomplete data was possible according to the methods defined in the study protocol and the SAP. No statistical analysis was performed.
Time Frame: Up to 10 weeks after first dose
Population: Randomised Set: All randomised subjects. Only 7 subjects were randomised into the study; 2 subjects completed the study as planned; therefore, no statistical analysis was performed.
  Due to low recruitment rate, the study was terminated early for non-safety reasons.
Measure: Mean (Full Range); unit: hours
Groups:
- CHF6563: Sublingual dose of CHF6563 and the corresponding oral dose of morphine matched placebo
  CHF6563
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
hours
  All treated patients | 157.62 [3.8 to 547.7] | 570.85 [501.5 to 640.2]
  Patients who completed the study (With Non Missing Data): number analyzed (Participants) | 1 | 1
  Patients who completed the study (With Non Missing Data) | 547.7 [547.7 to 547.7] | 501.5 [501.5 to 501.5]

2. Secondary Outcome: Time to First Weaning
Description: Record the time to first weaning, defined as the number of hours from first dose of study drug administration until the first dose reduction.
  The number of subjects randomised in the study was much lower than planned. Although data from 5 subjects were used in the CHF6563 treatment group, only 2 subjects completed the study as planned i.e. 1 subject in each study arm; no imputation of missing or incomplete data was possible according to the methods defined in the study protocol and the SAP. No statistical analysis was performed.
Time Frame: up to 10 weeks after first dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
hours
  All Treated Patients | 120.3 [120.3 to 120.3] | 56.2 [40.4 to 72.0]
  Patients who completed the study (With Non Missing Data): number analyzed (Participants) | 1 | 1
  Patients who completed the study (With Non Missing Data) | 120.3 [120.3 to 120.3] | 72 [72 to 72]

3. Secondary Outcome: Adjunctive Therapy
Description: Record the requirement for adjunctive drug therapy (phenobarbital) for signs of NOWS, recorded as Yes/No.
  Overall, 1 subject in the CHF6563 group and zero subjects in the morphine were reported as having received adjunctive drug therapy with phenobarbital.
  The number of subjects randomised in the study was much lower than planned. No imputation of missing or incomplete data was made. No statistical analysis was performed.
  NOWS=Neonatal Opioid Withdrawal Syndrome
Time Frame: up to 10 weeks after first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

4. Secondary Outcome: Requirement for Rescue Doses (CHF6563 or Morphine)
Description: Requirement for rescue doses and number of rescue doses administered (CHF6563 or morphine); (yes/no).
  The number of subjects randomised in the study was lower than planned. No imputation of missing or incomplete data was made. No statistical analysis was performed.
Time Frame: up to 10 weeks after first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
Participants
  Requirement for rescue doses -- Yes | 4 | 2
  Requirement for rescue doses -- No | 1 | 0

5. Secondary Outcome: Number of Rescue Doses Administered
Description: Number of rescue doses administered.
  The number of subjects randomised in the study was much lower than planned. Although data from 5 subjects were used in the CHF6563 treatment group, only 2 subjects completed the study as planned i.e. 1 subject in each study arm; no imputation of missing or incomplete data was possible according to the methods defined in the study protocol and the SAP. No statistical analysis was performed.
  At the discretion of the physician, a rescue dose of CHF6563 or morphine could be given during the up-titration phase or during the weaning phases to a neonate who had a single FNAST score ≥12. A rescue dose was not to be administered within 1 hour of the previous dose or 1 hour before the next scheduled dose. Rescue doses were the same as the previous dose.
Time Frame: up to 10 weeks after first dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: number of rescue doses
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
number of rescue doses
  All Treated Patients | 1.6 [0 to 4] | 3 [1 to 5]
  Patients who completed the study (With Non Missing Data): number analyzed (Participants) | 1 | 1
  Patients who completed the study (With Non Missing Data) | 4 [4 to 4] | 1 [1 to 1]

6. Secondary Outcome: Length of Opioid-related Hospital Stay
Description: Length of opioid-related hospital stay was defined as number of days from day of birth until 48 hours after the final dose of drug treatment for NOWS.
  Reported data show the length of opioid-related hospital stay (defined as number of days from day of birth until 48 hours after the final dose of drug treatment for NOWS).
  The number of subjects randomised in the study was much lower than planned. Although data from 5 subjects were used in the CHF6563 treatment group, only 2 subjects completed the study as planned i.e. 1 subject in each study arm; no imputation of missing or incomplete data was possible according to the methods defined in the study protocol and the SAP. No statistical analysis was performed.
Time Frame: up to 10 weeks plus 48 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: days
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
days
  All Treated Patients | 10.64 [3.9 to 27.0] | 29.5 [26.2 to 32.8]
  Patients who completed the study (With Non Missing Data): number analyzed (Participants) | 1 | 1
  Patients who completed the study (With Non Missing Data) | 27.0 [27.0 to 27.0] | 26.2 [26.2 to 26.2]

7. Secondary Outcome: Relapse of NOWS
Description: Relapse of NOWS, defined as experiencing recurrence of significant signs of withdrawal .
  Reported are subjects with experiencing a relapse.
  The number of subjects randomised in the study was much lower than planned. No imputation of missing or incomplete data was made. No statistical analysis was performed.
  NOWS=Neonatal Opioid Withdrawal Syndrome
Time Frame: up to 6 weeks after last dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF6563 | Morphine
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs and serious AEs (SAEs) were collected from the time of informed consent signature or from the neonate's birth through treatment and follow-up (FU) period (48 h after last treatment). Daily phone calls with the primary caregiver was for the first 7 d; weekly phone contact was up to 6 weeks after the final opioid treatment dose. NOWS treatment duration depends on Finnegan Neonatal Abstinence Scoring Tool (FNAST) scores and differs for each neonate; the maximum length of treatment was 10 weeks.
Description: Pre-treatment AEs=From between informed consent and first study drug administration. Treatment-emergent adverse events (TEAE)=From on or after first administration of any study drug. Peri-dosing AEs=AEs occurring during or shortly after (i.e., within 10 minutes) administration of study drug. Post-treatment AEs=From on or after the start of the FU phase (i.e. >48h after end of treatment). Ongoing AEs/SAEs were followed until the event resolved/stabilized, as acceptable to the Investigator.
Groups:
- CHF6563: Sublingual dose of CHF6563 and the corresponding oral dose of morphine matched placebo
  CHF6563: Sublingual CHF6563 administration at starting dose of 10 µg/kg q8
  Morphine matched-placebo: Oral morphine-matched placebo administration
- Morphine: Oral dose of morphine and the corresponding sublingual dose of CHF6563 matched placebo.
  Morphine: Oral morphine administration at starting dose of 0.07 mg/kg q4
  CHF6563 matched-placebo: Sublingual CHF6563 matched-placebo administration
Arm/Group | CHF6563 | Morphine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 2/5 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF6563 (N=5) | Morphine (N=2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poor feeding infant (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infantile vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Post-treatment AE
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Post-treatment AE

LIMITATIONS AND CAVEATS:
The study objectives could not be addressed because the study was terminated due to a low recruitment; for non-safety reasons.

Despite concerted efforts by the Sponsor to improve the enrolment rate (e.g., through communications with the Investigators, changing the training modalities to meet nurses' requests, and decreasing the sample size), the projected time frame to complete the study was longer than 5 years; this was considered unacceptable for the clinical development programme.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT04104646/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT04104646/SAP_001.pdf